CLINICAL TRIAL: NCT06265129
Title: The Association Between Obstructive Sleep Apnea Severity and Red Blood Cells Indices
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tamer Awad, Principal Investigator, Mansoura University
Other Study IDs: R.23.12.2429
Record Dates: First submitted 2024-02-10; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Erythrocyte Count; Erythrocyte Indices

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Complete blood picture (done in the morning after the night of monitored sleep by PSG. With stress on red blood cell indices (RBC count, MCV, MCH, RDW) — morning after the night of monitored sleep by PSG. With stress on red blood cell indices (RBC count, MCV, MCH, RDW)

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is characterized by recurrent episodes of obstructive events (apnea and hypopnea) and intermittent hypoxia, which in turn contributes to the systemic inflammation that underlies this disease and its consequences (Ryan et al 2009, Gileles-Hillel et al 2014). This systemic inflammation leads to endothelial dysfunction, which contributes to the pathogenesis of cardiovascular complications in OSAS, in addition to the exposure to risk factors, such as male gender, older age, obesity, and lack of exercise (Lorenzi Filho et al 2010). Some red blood cells (RBC) and platelets indices have emerged as inflammatory biomarkers in various diseases (Tertemiz et al 2016) The severity of OSA is significantly associated with increase hematocrit, even after controlling for possible confounding variables. However, nocturnal hypoxemia in OSA does not usually lead to clinical polycythemia (Choi et al 2006). In patients referred with a clinical diagnosis of OSAS, RDW may be a marker for the severity of the condition. As RDW is usually included in a complete blood count, it could provide an inexpensive tool for triaging OSAS patients for polysomnography evaluation (Sökücü et al 2012). The hematological indices white blood cell count (WBC), neutrophil count, lymphocyte count, mean platelet volume (MPV), platelet distribution width (PDW), and red blood cell distribution width (RDW) have been proposed as alternative markers to those normally used clinically, e.g., interleukin-6 (IL6) and C-reactive protein, to evaluate the burden of inflammation in OSAS (Wu et al 2018)

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is characterized by recurrent episodes of obstructive events (apnea and hypopnea) and intermittent hypoxia, which in turn contributes to the systemic inflammation that underlies this disease and its consequences (Ryan et al 2009, Gileles-Hillel et al 2014). This systemic inflammation leads to endothelial dysfunction, which contributes to the pathogenesis of cardiovascular complications in OSAS, in addition to the exposure to risk factors, such as male gender, older age, obesity, and lack of exercise (Lorenzi Filho et al 2010). Some red blood cells (RBC) and platelets indices have emerged as inflammatory biomarkers in various diseases (Tertemiz et al 2016) The severity of OSA is significantly associated with increase hematocrit, even after controlling for possible confounding variables. However, nocturnal hypoxemia in OSA does not usually lead to clinical polycythemia (Choi et al 2006). In patients referred with a clinical diagnosis of OSAS, RDW may be a marker for the severity of the condition. As RDW is usually included in a complete blood count, it could provide an inexpensive tool for triaging OSAS patients for polysomnography evaluation (Sökücü et al 2012). The hematological indices white blood cell count (WBC), neutrophil count, lymphocyte count, mean platelet volume (MPV), platelet distribution width (PDW), and red blood cell distribution width (RDW) have been proposed as alternative markers to those normally used clinically, e.g., interleukin-6 (IL6) and C-reactive protein, to evaluate the burden of inflammation in OSAS (Wu et al 2018)

Aim of Work:

To study the relationship between severity of obstructive sleep apnea and red blood cell indices

Study Design:

Retrospective Cross-sectional study

Patients and methods:

This cross-sectional study will be conducted at Chest Medicine Department, Sleep Disordered Breathing Unit, Mansoura university hospital on a thirty (30) patients with suspected obstructive sleep apnea (OSA)

Inclusion criteria:

1. Age above 18 years.
2. Stable patient with suspected OSA

Exclusion Criteria:

1. Age <18 years.
2. Pregnant females
3. Hemodynamically unstable patients
4. Patient with Chronic diseases like COPD, CHF, CKD, CLD. DM and Stroke
5. Patient with hematologic malignancies
6. Patient on anticoagulants
7. Patients with recent blood transfusion
8. Patient with psychosis Method

The patients enrolled in this study will be subjected to the following:

1. Full history taking and physical examination
2. OSA screening: ESS, Berlin questionnaire and STOP-Bang questionnaire,
3. Pulse oximetry
4. Full night attended polysomnography (PSG)
5. Laboratory Investigations:

   * Complete blood picture (done in the morning after the night of monitored sleep by PSG. With stress on red blood cell indices (RBC count, MCV, MCH, RDW)
   * Arterial blood gases if needed
   * Routine kidney function and liver function tests.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age above 18 years. 2. Stable patient with suspected OSA

Exclusion Criteria:

* 1. Age <18 years. 2. Pregnant females 3. Hemodynamically unstable patients 4. Patient with Chronic diseases like COPD, CHF, CKD, CLD. DM and Stroke 5. Patient with hematologic malignancies 6. Patient on anticoagulants 7. Patients with recent blood transfusion 8. Patient with psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: a thirty (30) patients with suspected obstructive sleep apnea (OSA)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Red Blood Cells Indices | one night
  Red Blood Cells Indices

CONTACTS AND LOCATIONS:
Locations (1):
- Tamer Awad Elsayed, Al Mansurah, Dakhlia, Egypt